CLINICAL TRIAL: NCT04530162
Title: Prevention of Post Herpetic Neuralgia by Ultrasound Guided Single Nerve Block in the Emergency Department
Brief Title: Prevention of Post Herpetic Neuralgia by Ultrasound Guided Single Nerve Block in the ED
Status: Withdrawn | Type: Observational
Why Stopped: No patients qualified for the study; PI left institution and current investigators lost interest in the study.
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 2019-09-04
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Pain
Keywords: pain; pain management; herpes zoster; ultrasound; emergency medicine
MeSH Terms: conditions — Pain; Agnosia; Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency Medicine Herpes Zoster Patients: Emergency Medicine adult patients with herpes zoster pain onset within 30 days of characteristic dermatomal herpes zoster rash who receive nerve block using bupivacaine and dexamethasone. The patient will be then started on Acyclovir 800 mg five times daily for seven days. For mild to moderate breakthrough pain, the patient will be prescribed a 5-day course of Tylenol 650 mg and Ibuprofen 400 mg taken up to every 8 hours together. For severe breakthrough pain, the patients will be prescribed a two-day course of 7.5 mg morphine sulfate immediate release to be taken up to every 6 hours. The location of the nerve block and dosage of injected medications will depend on the distribution of the affected dermatome.
  Interventions: Procedure: Ultrasound guided nerve block

INTERVENTIONS:
Procedure: Ultrasound guided nerve block — nerve block using bupivacaine and dexamethasone.

SUMMARY:
Herpes zoster causes significant morbidity on over 1 million Americans every year. Although the majority of herpes zoster pain will self-resolve within one week, a significant proportion of patients will develop postherpetic neuralgia (PHN), which is characterized by debilitating pain that persists more than three months after the initial symptoms. Nerve blocks have been previously studied as a method to control herpes zoster pain in outpatient pain clinics and inpatient settings. This study aims to investigate whether emergency department ultrasound guided nerve blocks can prevent PHN and effectively treat acute herpes zoster pain.

DETAILED DESCRIPTION:
Study Objectives The goal of this study is to evaluate the rate of PHN development in emergency department patients who receive ultrasound guided nerve blocks using bupivacaine and dexamethasone for acute herpes zoster. The investigators will also study the effectiveness of the block in managing acute herpes zoster pain. The primary outcome is the percentage of patients who have significant herpetic pain at 1 month and 3 months after receiving the nerve block. Secondary outcomes measured are pain scores at 1 hour, 1 month, and 3 months post-nerve block. The amount of opioids used after discharge as well as the number of return visits for herpetic pain will also be recorded.

Hypothesis The hypothesis is that patients who receive nerve blocks will decrease the occurrence of PHN development at 1 month and 3 months post-treatment. The secondary hypothesis is that nerve blocks will decrease pain scores at 1 hour, 1 month, 3 months, as well as reduce the amount of opioids used and number of return visits for herpetic pain.

IStudy Design This study will be a single center prospective observational study that will be conducted in the emergency department of an urban hospital center. A trained emergency medicine physician will screen and assess the patient for eligibility. Once the patient is determined to be eligible, informed consent will be obtained. A trained EM physician will then administer a nerve block using bupivacaine and dexamethasone to a patient with acute herpes zoster. The patient will be started on Acyclovir 800 mg five times daily for seven days. For mild to moderate breakthrough pain, the patient will be prescribed a 5-day course of Tylenol 650 mg and Ibuprofen 400 mg taken up to every 8 hours together. For severe breakthrough pain, the patients will be prescribed a two-day course of 7.5 mg morphine sulfate immediate release to be taken up to every 6 hours. The location of the nerve block and dosage of injected medications will depend on the distribution of the affected dermatome. The dermatomal distributions with their associated nerve blocks and medication dosages are shown the table below.

Herpes Zoster Distribution Nerve Block Type Medication T2-T9 Serratus Plane 30 mL 0.25% bupivacaine and 8 mg Dexamethasone C2-C3 Greater Occipital Nerve 2 mL 0.25% bupivacaine and 4 mg dexamethasone C3-C4 Superficial Cervical Plexus 10 mL 0.25% bupivacaine and 4 mg dexamethasone Anterior Abdominal Wall T6 - L1 Transversus Abdominis Plane 30 mL 0.25% bupivacaine and 8 mg dexamethasone

A numerical verbal rating scale will be used to assess the patient's pain pre-injection and at 1-hour post nerve block. We will then call the patient at the 1 week, 1 month, and 3-month post-nerve block time intervals to assess the patients' pain. The investigators will also record the number of follow-up visits for herpetic pain and the amount of additional pain medications used.

When called the patient will be asked a series of questions:

1. Do you continue to have pain associated with your herpes zoster infection?
2. If so, how would you rate your pain from a scale of 0-10? 10 being the worst pain you have ever had in your life.
3. About how much pain medication have you been using since the initial nerve block? How many doses of Ibuprofen or Tylenol per day for how many days? How many doses of morphine sulfate immediate release or other opioids were taken per day for how many days?
4. If you used other forms of pain controllers, what were they and how often and for how long did you use them?
5. Have you seen your primary care doctor, pain clinic, emergency department, or other pain management follow-up visits for management of your herpes pain? If so, how many visits have you made?
6. What side effects have you had since the nerve block?

Subjects:

The study population is Maimonides Medical Center emergency department patients older than 18 years of age presenting with acute herpes zoster patient with characteristic dermatomal vesicular skin lesions within 30 days of initial symptoms.

Design:

The primary outcome is the percentage of patients who have significant herpetic pain at 1 month and 3 months after receiving the nerve block. Secondary outcomes measured are pain scores pre-injection, and 1 hour, 1 month, and 3 months post-nerve block. The number of tablets of opioids and other analgesics used after discharge as well as the number of return visits for herpetic pain will also be recorded.

Data Collection Procedures:

The numerical verbal rating scale pain score will be recorded by a research staff member at 1 hour after administration of nerve block. The patients will then be called at 1 week, 1 month, and 3 months post nerve block for assessment of NRS as well as number of follow-up visits and amount of analgesics used. A medication track form/log will be given to the patients to help record the amount of medications taken in the first week. The patients will be stratified by age: those under 50, 50-59, 60-69, and 70 and older as well as herpes zoster vaccination status.

Expected Outcomes:

The investigators expect that patients undergoing ultrasound guided nerve block will have decreased incidence of subacute herpetic neuralgia and PHN. We also expect pain to be well controlled at 1 hour, 1 week, 1 month, and 3 months post nerve block.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18
2. herpes zoster pain
3. pain onset within 30 days of characteristic dermatomal herpes zoster rash

Exclusion Criteria:

1. allergic to bupivacaine
2. signs of infection over herpes zoster site
3. greater than 30 days duration of pain
4. pain across more than one dermatome
5. pregnant and/or breastfeeding

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is Maimonides Medical Center emergency department patients older than 18 years of age presenting with acute herpes zoster patient with characteristic dermatomal vesicular skin lesions within 30 days of initial symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence of subacute herpetic neuralgia | 1 month
  The number of new cases of subacute herpetic neuralgia

SECONDARY OUTCOMES:
Pain Control | 1 month
  Pain score on an 11 point Likert scale ranging from 0 to 10 where 0 is no pain, 5 is moderate pain and 10 is very severe pain.

OTHER OUTCOMES:
Incidence of post herpetic neuralgia | 1 month
  The number of new cases of post herpetic neuralgia

CONTACTS AND LOCATIONS:
Overall Officials: Leily Naraghi, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT04530162/Prot_001.pdf